CLINICAL TRIAL: NCT06166251
Title: Effects of a Single Bout of Low and Moderate Intensity Aerobic Exercise on Acquisition and Retention of Motor Learning in Young Adults
Brief Title: The Effects of Exercise Timing and Intensity on Motor Learning in Healthy Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Muhammed Şeref Yıldırım, Research Assistant (PhD), Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TU-FTR-MŞY-001
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: exercise; motor skills; retention; Young Adult; Sleep Quality
MeSH Terms: conditions — Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: 75 young adults were divided into five groups: two groups that did low or moderate intensity aerobic exercise before motor practice (LOW-MP, MOD-MP), two groups that did aerobic exercise after motor practice (MP-LOW, MP-MOD), and non-exercise control group.
Who Masked: Participant
Masking Description: Participants were not informed that there were different intensity and timing groups. In addition, the participant did not know whether he/she was exercising at moderate or low intensity because the speed of the treadmill during the exercise was adjusted by the therapist according to a predetermined target heart rate.
  The participant's heart rate was monitored with a polar heart rate monitor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MP-LOW (pre-motor practice (MP) low ıntensity aerobic exercise ) (Experimental): On the experimental day, they participated in 60 golf puttings (acquisition practice) followed by a half-hour low-intensity treadmill run.
  Retention levels were measured 1 and 7 days after the experimental day with 10 puttings each.
  Sleep quality (richard campbell sleep questionnaire) and cognitive level (Paced auditory serial addition test) were evaluated in all participants.
  Interventions: Behavioral: low ıntensity aerobic exercise
- MP-MOD (pre-motor practice (MP) moderate ıntensity aerobic exercise ) (Experimental): On the experimental day, they participated in 60 golf puttings (acquisition practice) followed by a half-hour moderate-intensity treadmill run.
  Retention levels were measured 1 and 7 days after the experimental day with 10 puttings each.
  Sleep quality (richard campbell sleep questionnaire) and cognitive level (Paced auditory serial addition test) were evaluated in all participants.
  Interventions: Behavioral: moderate ıntensity aerobic exercise
- MOD-MP (post-motor practice (MP) moderate ıntensity aerobic exercise ) (Experimental): On the experimental day, they participated in a half-hour moderate-intensity treadmill run followed by 60 golf puttings (acquisition practices).
  Retention levels were measured 1 and 7 days after the experimental day with 10 puttings each.
  Sleep quality (richard campbell sleep questionnaire) and cognitive level (Paced auditory serial addition test) were evaluated in all participants.
  Interventions: Behavioral: moderate ıntensity aerobic exercise
- LOW-MP ((post-motor practice (MP) low ıntensity aerobic exercise ) (Experimental): On the experimental day, they participated in a half-hour low-intensity treadmill run followed by 60 golf puttings (acquisition practices).
  Retention levels were measured 1 and 7 days after the experimental day with 10 puttings each.
  Sleep quality (richard campbell sleep questionnaire) and cognitive level (Paced auditory serial addition test) were evaluated in all participants.
  Interventions: Behavioral: low ıntensity aerobic exercise
- Control (No Intervention): On the experimental day, they completed 60 golf puttings (just acquisition practices- NO EXERCISE) Retention levels were measured 1 and 7 days after the experimental day with 10 puttings each.
  Sleep quality (richard campbell sleep questionnaire) and cognitive level (Paced auditory serial addition test) were evaluated in all participants.

INTERVENTIONS:
Behavioral: low ıntensity aerobic exercise — The exercise intervention was 30 min of treadmill jogging/running. After a two-minute warm-up walk at 1.0 m/s, the treadmill speed was increased to 57-63% maximum heart rate.
  Arms: LOW-MP ((post-motor practice (MP) low ıntensity aerobic exercise ); MP-LOW (pre-motor practice (MP) low ıntensity aerobic exercise )
Behavioral: moderate ıntensity aerobic exercise — The exercise intervention was 30 min of treadmill jogging/running. After a two-minute warm-up walk at 1.0 m/s, the treadmill speed was increased to 64-76% maximum heart rate.
  Arms: MOD-MP (post-motor practice (MP) moderate ıntensity aerobic exercise ); MP-MOD (pre-motor practice (MP) moderate ıntensity aerobic exercise )

SUMMARY:
The purpose of this study is to compare of the effects of a single session of aerobic exercise with different intensity and timing on motor learning processes in healthy young adults.

DETAILED DESCRIPTION:
Long-term aerobic training are associated with improved motor learning. Recent studies have shown that even a single bout of moderate or high ıntensity aerobic exercise can lead to immediate improvements on motor learning. On the other hand, there is still insufficient knowledge about whether aerobic exercise should occur before or after motor practice and what the intensity of aerobic exercise should be. In this study, the ınvestigators examined the effects of a single bout of low and moderate intensity aerobic exercise applied before or after motor practice on golf putting task. Additionally, the ınvestıgators evaluated the effects of sleep quality on motor learning and the acute effects of the exercise on cognition. 75 young adults were divided into five groups: two groups that did low or moderate intensity aerobic exercise before motor practice (LOW-MP, MOD-MP), two groups that did aerobic exercise after motor practice (MP-LOW, MP-MOD), and non-exercise control group. The acquisition practice consisted of six blocks of ten golf puttings. The retention was also evaluated both 1 day and 7 days after the experimental day with one block each. The putting performance was measured with accuracy and consistency error scores were computed for each acquisition and retention block. The sleep quality of the night before and the experimental day were evaluated using the Richard Campbell Sleep Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-24 years
* Risk score less than two based on The American Heart Association (AHA) and American College of Sports Medicine (ACSM) health/fitness facility pre-participation screening questionnaire
* Physical activity level>1500 MET/min weeks based on the International Physical Activity Questionnaire (IPAQ)

Exclusion Criteria:

* being elite athletes
* being smokers
* using psychiatric/neurologic medications.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Bivariate variable error score (BVE) | For each of 8 golf putting blocks (6 acquisition blocks on the experimental day, 1 retention block 1 day after the experimental day and 1 retention block 7 days after the experimental day
  The distance of the ball to the target in the x- and y-coordinates was recorded for each putting with the help of coordinate lines drawn on the artificial grass mat. Recorded coordinates were used to calculate the bivariate variable error (BVE) scores. The BVE, also referred to as consistency, was measured, as the average of the absolute distance to the subject's own midpoint. Each subject's midpoint was measured as the average hit location over ten puttings for each block. Lower BVE indicates greater consistency.
Median Radial Error (MRE) | For each of 8 golf putting blocks (6 acquisition blocks on the experimental day, 1 retention block 1 day after the experimental day and 1 retention block 7 days after the experimental day
  The distance of the ball to the target in the x- and y-coordinates was recorded for each putting with the help of coordinate lines drawn on the artificial grass mat. Recorded coordinates were used to calculate the Median Radial Error (MRE) scores. The mean radial error (MRE) was measured as the average of the absolute distances to the centre of the target of the 10 shots comprising each block.

SECONDARY OUTCOMES:
Paced auditory serial addition task (PASAT) | For the four exercise groups: On the experimental day 2 times immediately before and after the half-hour exercise For control group: immediately before and after the half-hour rest.
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and working memory, as well as calculation ability. The PASAT is presented using recording tape to ensure standardization in the rate of stimulus presentation. Single digits are presented every 2 seconds and the patient must add each new digit to the one immediately prior to it. The score for the PASAT is the total number correct out of 60 possible answers.
Richard Campbell Sleep Questionnaire (RCSQ) | Day 1 (experimental day) and Day 2 (1 day retention visit)
  The RCSQ is a five-item self-report questionnaire that is used in order to assess perceived sleep depth, sleep latency (time to fall asleep), and number of awakenings, as well as sleep efficiency and quality.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Ş Yıldırım, PhD, Principal Investigator — Trakya University
Locations (1):
- Faculty of Health Science, Trakya University, Edirne, İskender, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I can share my data with all participants who contact me by e-mail.